CLINICAL TRIAL: NCT02161575
Title: A Phase IV, Prospective, Open-label, Uncontrolled, European Study in Patients With Neovascular Age-related Macular Degeneration (nAMD), Evaluating the Efficacy and Safety of Switching From Intravitreal Aflibercept to Ranibizumab 0.5mg.
Brief Title: Safety and Efficacy of Switching From Aflibercept to Ranibizumab in Patients With nAMD
Acronym: SAFARI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002AGB17; 2014-001085-10 (EudraCT Number)
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Macular degeneration; age-related macular degeneration (ARMD); vision loss; macula damage; retina damage; dry macular degeneration; wet macular degeneration; AMD
MeSH Terms: conditions — Macular Degeneration; Vision Disorders; Geographic Atrophy; Wet Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ranibizumab (Experimental): All patients received 3 monthly intraveal injections of 0.5mg ranibizumab followed by monthly injections of ranibizumab 0.5mg for a further 3 months on a prn (as required) basis, as determined by the study doctor.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intraveal injections of 0.5mg ranibizumab

SUMMARY:
AMD (Age Related Macular Degeneration) is the leading cause of severe visual loss and blindness registration in the UK . It is a disease which affects the retina (the nerve and blood vessel network at the back of the eye responsible for vision). Patients can suffer with severe visual loss and have difficulties with every day tasks such as recognising faces, reading & driving.

There are two variations of the disease, a 'dry' type & a 'wet' type also known as neovascular AMD (nAMD). In wet/nAMD new vessels grow from the blood supply underneath the retina, in part due to higher than normal levels of a protein called Vascular Endothelial Growth Factor (VEGF). Since the introduction of drugs which block VEGF, visual outcomes for patients with wAMD have dramatically improved.

There are 2 widely used treatments; ranibizumab and aflibercept. Whilst the majority of patients have a successful outcome with treatment, many patients experience suboptimal response. This study evaluated if these patients experience a benefit from a switch to a different antiVEGF drug treatment.

In this study nAMD patients who are showing no or poor to response to treatment with aflibercept were switched to ranibizumab to assess if there is any benefit in terms of treatment outcomes.

Patients visited the hospital clinic 8 times over the 7 - 8 month study period. Monthly ranibizumab injections were given for the first 3 months, then monthly as required for the next 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity (BCVA) ≥23 ETDRS letters in study eye
* Evidence of active choroidal neovascularisation (CNV) involving the center of the fovea in study eye Patient subgroup specific inclusion criteria: - Group 1. Primary treatment failure
* Initiated treatment with aflibercept <130 days prior to the Screening Visit.
* No increase in BCVA (≥5 letters) since commencing treatment with aflibercept.
* Disease activity has never been controlled in the study eye after initiating aflibercept as defined by at least one of the following: evidence of unchanged or increasing retinal or subretinal fluid; new PED; unchanged or increasing size of preexisting PED.

Group 2. Suboptimal treatment response

* Aflibercept commenced ≥6 months prior to the Screening Visit.
* Received ≥3 aflibercept injections into the study eye within 6 months of the Screening Visit.
* Evidence of previous reduced disease activity (as defined by reduction of ≥50μm in Central Subfield Retinal Thickness on OCT) noted in the study eye after initiating aflibercept.
* At Screening Visit, disease activity has worsened (as defined by increasing retinal* or subretinal fluid, or new or increasing size of PED) in the study eye compared to prior visits.

Exclusion Criteria:

* History of cerebrovascular accident, transient ischemic attack or myocardial infarction within 3 months of the Screening visit.
* Uncontrolled blood pressure
* Evidence of bilateral active CNV during the Screening Period or at Baseline requiring bilateral antiVEGF injections.
* Prior intravitreal injection of ranibizumab or bevacizumab into the study eye and/or prior intravitreal injection of bevacizumab into the fellow eye.
* Cataract (if causing significant visual impairment), aphakia, severe vitreous hemorrhage, rhegmatogenous retinal detachment, proliferative retinopathy or choroidal neovascularization of any other cause than wet AMD (e.g. ocular histoplasmosis, pathologic myopia (≥8 dioptres)) at the time of Screening and Baseline.
* Irreversible structural damage involving the center of the fovea (e.g. advanced fibrosis or geographic atrophy) which in the opinion of the Investigator is sufficient to irreversibly impair visual acuity.
* Polypoidal choroidal vasculopathy (PCV), RPE tear, central serous retinopathy (CSR), or significant vitreomacular traction identified during Screening period or within 4 months of Baseline visit.
* Unable to obtain at Screening OCT images of sufficient quality to be analyzed

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (26):
- Germany (6):
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mühlheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
- United Kingdom (20):
  - Novartis Investigative Site, Darlington, Durham
  - Novartis Investigative Site, Harlow, Essex
  - Novartis Investigative Site, Canterbury, Kent
  - Novartis Investigative Site, Aberdeen, Scotland
  - Novartis Investigative Site, Ipswich, Suffolk
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, East Kilbride
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Great Yarmouth
  - Novartis Investigative Site, Harrogate
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Sunderland
  - Novartis Investigative Site, Uxbridge
  - Novartis Investigative Site, York

REFERENCES:
- [Derived] Gale RP, Pearce I, Eter N, Ghanchi F, Holz FG, Schmitz-Valckenberg S, Balaskas K, Burton BJL, Downes SM, Eleftheriadis H, George S, Gilmour D, Hamilton R, Lotery AJ, Patel N, Prakash P, Santiago C, Thomas S, Varma D, Walters G, Williams M, Wolf A, Zakri RH, Igwe F, Ayan F. Anatomical and functional outcomes following switching from aflibercept to ranibizumab in neovascular age-related macular degeneration in Europe: SAFARI study. Br J Ophthalmol. 2020 Apr;104(4):493-499. doi: 10.1136/bjophthalmol-2019-314251. Epub 2019 Aug 5. PMID 31383649

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 22 sites located in the United Kingdom and 6 sites located in Germany. A total of 103 patients received at least 1 dose of study drug.
Pre-assignment Details: Of the 103 patients who received at least 1 dose of study drug, 3 patients did not have any post-baseline safety or CSRT assessments and were therefore excluded from the SAF and FAS, in accordance with the analysis set definitions. Therefore, 100 patients were included in the SAF and FAS.
Period: Overall Study
Arm/Group | Ranibizumab
Started | 103
Full Analysis Set (FAS) Population (received an application of study treatment and had a baseline and post-baseline assessment for CSRT) | 100
Safety (SAF) Population (received an application of study treatment and and had at least one post-baseline safety assessment) | 100
Completed | 92
Not Completed | 11
Not completed — Protocol Violation | 8
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: FAS
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: FAS
  years | 77 (6.51)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Female | 55
    Male | 45
Race/Ethnicity, Customized [Number; unit: Participants] — Population: FAS
  Participants
    Caucasian | 99
    Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Central Subfield Retinal Thickness (CSRT) From Baseline to Day 90.
Description: Measurement of the change in CSRT, determined by high definition optical coherence tomography (HD-OCT) after 3 monthly injections of ranibizumab. OCT is a non-invasive technique which can determine and measure thickness of the retina. A negative change from Baseline indicates an improvement (less retinal fluid and lower disease activity). Data collected on the study eye were used for the evaluation of efficacy.
Time Frame: Baseline and Day 90
Population: FAS - Missing values at Day 90 were imputed using Last Observation Carried Forward (LOCF) where possible. For the change from baseline, only patients with a value at both baseline and Day 90 were included.
Measure: Median (Full Range); unit: micrometer
Arm/Group | Ranibizumab
Number analyzed (Participants) | 97
micrometer
  Baseline | 384.00 [154.0 to 975.0]
  Day 90 | 318.00 [170.0 to 832.0]
  Change from Baseline to Day 90: number analyzed (Participants) | 94
  Change from Baseline to Day 90 | -30.75 [-386.0 to 78.0]
Statistical Analysis 1: Comparison: Ranibizumab; The null hypothesis was that the change in CSRT from baseline to Day 90 was zero; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Confidence Interval for the Median Change form Baseline; Median Difference (Final Values) = -30.75, 95% CI 2-sided [-59.50 to -20.50]

2. Secondary Outcome: Change in Subfoveal Retinal Thickness (SRT) From Baseline to Day 180
Description: Measurement of change in SRT from Baseline to Day 180 as determined by high definition optical coherence tomography (HD-OCT). A reduction indicates an improvement in overall disease activity. Data collected on the study eye were used for the evaluation of efficacy.
Time Frame: Baseline and Day 180
Population: FAS
Measure: Median (Full Range); unit: micrometer
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
micrometer
  SRT at Baseline | 346.00 [69.0 to 944.5]
  SRT at Day 180: number analyzed (Participants) | 93
  SRT at Day 180 | 302.00 [41.5 to 876.5]
  SRT change from Baseline to Day 180: number analyzed (Participants) | 93
  SRT change from Baseline to Day 180 | -23.50 [-464.0 to 306.5]

3. Secondary Outcome: Change in Central Subfield Retinal Thickness (CSRT) From Baseline to Day 180
Description: Measurement of change in CSRT from Baseline to Day 180 as determined by high definition optical coherence tomography (HD-OCT). A reduction indicates an improvement in overall disease activity. Data collected on the study eye were used for the evaluation of efficacy.
Time Frame: Baseline and Day 180
Population: FAS
Measure: Median (Full Range); unit: micrometer
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
micrometer
  CSRT at Baseline: number analyzed (Participants) | 97
  CSRT at Baseline | 384.00 [154.0 to 975.0]
  CSRT at Day 180: number analyzed (Participants) | 88
  CSRT at Day 180 | 343.00 [194.0 to 842.0]
  CSRT change from Baseline to Day 180: number analyzed (Participants) | 85
  CSRT change from Baseline to Day 180 | -28.00 [-271.0 to 171.0]

4. Secondary Outcome: Change in Central Subfield Retinal Volume (CSRV) From Baseline to Day 180
Description: Measurement of change in CSRV from Baseline to Day 180 as determined by high definition optical coherence tomography (HD-OCT). A reduction indicates an improvement in overall disease activity. Data collected on the study eye were used for the evaluation of efficacy.
Time Frame: Baseline and Day 180
Population: FAS
Measure: Median (Full Range); unit: cubic micrometer
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
cubic micrometer
  CSRV at Baseline: number analyzed (Participants) | 90
  CSRV at Baseline | 0.3050 [0.120 to 11.600]
  CSRV at Day 180: number analyzed (Participants) | 76
  CSRV at Day 180 | 0.2750 [0.115 to 11.400]
  CSRV change from Baseline to Day 180: number analyzed (Participants) | 74
  CSRV change from Baseline to Day 180 | -0.0200 [-1.600 to 0.135]

5. Secondary Outcome: Number of Patients With Intraretinal Fluid Assessed at Baseline and Day 180
Description: Presence or absence of qualitative OCT parameter Intraretinal Fluid. Data collected on the study eye were used for the evaluation of efficacy.
Time Frame: Baseline and Day 180
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
Participants
  Baseline: Yes, Definitive | 32
  Baseline: Yes, Subtle | 11
  Baseline: No | 56
  Baseline: Questionable | 1
  Day 180: number analyzed (Participants) | 94
  Day 180: Yes, Definitive | 24
  Day 180: Yes, Subtle | 15
  Day 180: No | 55
  Day 180: Questionable | 0

6. Secondary Outcome: Number of Patients With Subretinal Fluid Assessed at Baseline and Day 180
Description: Presence or absence of qualitative OCT parameter Subretinal Fluid. Data collected on the study eye were used for the evaluation of efficacy.
Time Frame: Baseline to Day 180
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
Participants
  Baseline: Yes, Definitive | 83
  Baseline: Yes, Subtle | 5
  Baseline: No | 12
  Day 180: number analyzed (Participants) | 94
  Day 180: Yes, Definitive | 49
  Day 180: Yes, Subtle | 15
  Day 180: No | 30

7. Secondary Outcome: Number of Patients With Intraretinal/Subretinal Fluid Within the Central Subfield Fluid Assessed at Baseline and Day 180
Description: Presence or absence of qualitative OCT parameter Intraretinal/Subretinal Fluid Within the Central Subfield. Data collected on the study eye were used for the evaluation of efficacy.
Time Frame: Baseline and Day 180
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
Participants
  Baseline: Yes, Definitive | 38
  Baseline: Yes, Subtle | 6
  Baseline: No | 5
  Baseline: Questionable | 1
  Baseline: NA | 50
  Day 180: number analyzed (Participants) | 94
  Day 180: Yes, Definitive | 26
  Day 180: Yes, Subtle | 12
  Day 180: No | 15
  Day 180: Questionable | 1
  Day 180: NA | 40

8. Secondary Outcome: Number of Patients With Pigment Epithelial Detachments Assessed at Baseline and Day 180
Description: Presence or absence of qualitative OCT parameter Pigment Epithelial Detachments. Data collected on the study eye were used for the evaluation of efficacy.
Time Frame: Baseline and Day 180
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
Participants
  Baseline: Yes, Definitive | 86
  Baseline: Yes, Subtle | 2
  Baseline: No | 12
  Baseline: Not gradable | 0
  Day 180: number analyzed (Participants) | 94
  Day 180: Yes, Definitive | 80
  Day 180: Yes, Subtle | 4
  Day 180: No | 8
  Day 180: Not gradable | 2

9. Secondary Outcome: Number of Patients With Dry Retina Assessed at Baseline and Day 180
Description: Presence or absence of qualitative OCT parameter Dry Retina. Data collected on the study eye were used for the evaluation of efficacy.
Time Frame: Baseline and Day 180
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
Participants
  Baseline: Yes, Definitive | 0
  Baseline: No | 100
  Day 180: number analyzed (Participants) | 94
  Day 180: Yes, Definitive | 0
  Day 180: No | 94

10. Secondary Outcome: Change in Maximum PED Height From Baseline to Day 180
Description: Change from Baseline to Day 180 in Maximum Pigment Epithelial Detachment (PED) Height. Data collected on the study eye were used for the evaluation of efficacy.
Time Frame: Baseline and Day 180
Population: FAS
Measure: Median (Full Range); unit: micrometer
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
micrometer
  Baseline: number analyzed (Participants) | 93
  Baseline | 236.00 [66.5 to 674.0]
  Day 180: number analyzed (Participants) | 83
  Day 180 | 203.50 [63.5 to 705.0]
  Change from Baseline to Day 180: number analyzed (Participants) | 80
  Change from Baseline to Day 180 | -2.50 [-336.5 to 131.0]

11. Secondary Outcome: Change in Maximum PED Diameter From Baseline to Day 180
Description: Change from Baseline to Day 180 in Maximum Pigment Epithelial Detachment (PED) Diameter. Data collected on the study eye were used for the evaluation of efficacy.
Time Frame: Baseline and Day 180
Population: FAS
Measure: Median (Full Range); unit: micrometer
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
micrometer
  Baseline: number analyzed (Participants) | 93
  Baseline | 2205.00 [0.0 to 4877.0]
  Day 180: number analyzed (Participants) | 83
  Day 180 | 2428.00 [471.0 to 4683.0]
  Change from Baseline to Day 180: number analyzed (Participants) | 80
  Change from Baseline to Day 180 | 59.50 [-1007.0 to 2756.0]

12. Secondary Outcome: Change in Maximum IRC Height From Baseline to Day 180
Description: Change from Baseline to Day 180 in Maximum Intraretinal Cyst (IRC) Height. Data collected on the study eye were used for the evaluation of efficacy.
Time Frame: Baseline and Day 180
Population: FAS
Measure: Median (Full Range); unit: micrometer
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
micrometer
  Baseline: number analyzed (Participants) | 42
  Baseline | 121.50 [21.0 to 280.5]
  Day 180: number analyzed (Participants) | 33
  Day 180 | 105.50 [25.5 to 485.0]
  Change from Baseline to Day 180: number analyzed (Participants) | 29
  Change from Baseline to Day 180 | 0.00 [-223.5 to 235.0]

13. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA was assessed as letters read and measured in a sitting position using subjective refraction and Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at an initial testing distance of 4 meters.
Time Frame: Baseline, Day 90 and Day 180
Population: FAS
Measure: Median (Full Range); unit: letters
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
letters
  Baseline | 71.5 [36 to 90]
  Day 90: number analyzed (Participants) | 94
  Day 90 | 74.0 [32 to 87]
  Day 180: number analyzed (Participants) | 97
  Day 180 | 75.0 [32 to 90]
  Change from Baseline to Day 180: number analyzed (Participants) | 97
  Change from Baseline to Day 180 | 1.0 [-31 to 35]
  Change from Day 90 to Day 180: number analyzed (Participants) | 92
  Change from Day 90 to Day 180 | 0.0 [-25 to 24]

14. Secondary Outcome: Change in ETDRS Letters for Study Eye From Baseline to Day 180
Description: Number of patients gaining at least 15 letters from Baseline to Day 180
Time Frame: Baseline and Day 180
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
Participants
  >=15 (Gain of at least 15 letters) | 11
  10 to <15 | 6
  5 to <10 | 17
  0 to <5 | 25
  >-15 to <0 | 31
  <=-15 (Loss of at least 15 letters) | 7
  NA | 3

15. Secondary Outcome: Incidence of Ocular TEAEs in the Study Eye Reported by ≥2% Patients From Baseline to Day 180
Description: Incidence of ocular Treatment Emergent Adverse Events (TEAEs) in the study eye reported by ≥2% patients by preferred term.
Time Frame: Baseline to Day 180
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 100
Participants
  Eye pain | 3
  Visual impairment | 3
  Blepharitis | 2
  Posterior capsule opacification | 2
  Intraocular pressure increased | 3

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 6 months.
Description: Ocular AEs are reported for the study eye and non-study eye combined.
Arm/Group | Ranibizumab
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 10/100
Other Adverse Events (participants affected / at risk) | 52/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=100)
ANAEMIA (Blood and lymphatic system disorders) | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1
ATRIAL FLUTTER (Cardiac disorders) | 1
RETINAL HAEMORRHAGE (Eye disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1
PNEUMONIA (Infections and infestations) | 1
CONTUSION (Injury, poisoning and procedural complications) | 1
FALL (Injury, poisoning and procedural complications) | 3
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1
CATHETERISATION CARDIAC (Investigations) | 1
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 1
PROSTATOMEGALY (Reproductive system and breast disorders) | 1
UMBILICAL HERNIA REPAIR (Surgical and medical procedures) | 1
VAGINAL PROLAPSE REPAIR (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.9% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=100)
ANAEMIA (Blood and lymphatic system disorders) | 2
BLEPHARITIS (Eye disorders) | 6
DRY EYE (Eye disorders) | 3
EYE PAIN (Eye disorders) | 3
POSTERIOR CAPSULE OPACIFICATION (Eye disorders) | 2
VISUAL IMPAIRMENT (Eye disorders) | 3
FATIGUE (General disorders) | 2
CYSTITIS (Infections and infestations) | 2
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7
NASOPHARYNGITIS (Infections and infestations) | 9
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
BLOOD PRESSURE INCREASED (Investigations) | 4
BLOOD PRESSURE SYSTOLIC INCREASED (Investigations) | 2
HEART RATE DECREASED (Investigations) | 2
INTRAOCULAR PRESSURE INCREASED (Investigations) | 3
WEIGHT DECREASED (Investigations) | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2
DIZZINESS (Nervous system disorders) | 2
HEADACHE (Nervous system disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 7
HYPERTENSION (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT02161575/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT02161575/SAP_001.pdf